CLINICAL TRIAL: NCT00829426
Title: A Relative Bioavailability Study of 3 mg Alprazolam Extended Release Tablets Under Fasting Conditions
Brief Title: Alprazolam Extended-Release 3mg Tablets Bioequivalence Study Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: R05-0166
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Results first posted 2009-07-21 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Alprazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alprazolam (Experimental): Alprazolam 3mg ER Tablet (test) dosed in first period followed by Xanax XR® 3 mg Tablet (reference) dosed in second period
  Interventions: Drug: Alprazolam Extended-Release 3 mg Tablets
- Xanax XR® (Active Comparator): Xanax XR® 3 mg Tablet (reference) dosed in first period followed by Alprazolam 3 mg ER Tablet (test) dosed in second period
  Interventions: Drug: Alprazolam Extended-Release 3 mg Tablets

INTERVENTIONS:
Drug: Alprazolam Extended-Release 3 mg Tablets — 1 x 3 mg, single dose fasting
  Arms: Alprazolam
Drug: Alprazolam Extended-Release 3 mg Tablets — 1 x 3 mg, single dose fasting
  Other Names: XANAX XR®
  Arms: Xanax XR®

SUMMARY:
This study will compare the relative bioavailability (rate and extent of absorption) of 3 mg Alprazolam Extended Release Tablets manufactured and distributed by TEVA Pharmaceuticals USA with that of 3 mg XANAX XR® Tablets by Pharmacia & Upjohn Company following a single oral dose (1 x 3 mg extended release tablet) in healthy adult subjects administered under fasting conditions.

DETAILED DESCRIPTION:
Detailed Description

Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

Outcome: Confidence interval fell within 80-125% therefore met the FDA Bioequivalence criteria; no drug related, serious, unexpected adverse events were reported during the study.

ELIGIBILITY:
Inclusion Criteria:

* Screening Demographics: All subjects selected for this study will be healthy non-smoking men and women 18 years of age or older at the time of dosing. The subject's body mass index (BMI) should be less than or equal to 30.
* Screening procedures: Each subject will complete the screening process within 28 days prior to Period I dosing.
* Consent documents for both the screening evaluation and HIV antibody determination will be reviewed, discussed, and signed by each potential participant before full implementation of screening procedures.
* Screening will include general observations, physical examination, demographics, medical and medication history, an electrocardiogram, sitting blood pressure and heart rate, respiratory rate and temperature.
* The physical examination will include, but may not be limited to an evaluation of the cardiovascular, gastrointestinal, respiratory, and central nervous systems.
* The screening clinical laboratory procedures will include:

  * Hematology: hematocrit, hemoglobin, WBC count with differential, RBC count, platelet count;
  * Clinical Chemistry: serum creatinine, BUN, glucose, AST(GOT), ALT(GPT), albumin, total bilirubin, total protein, and alkaline phosphatase;
  * HIV antibody, hepatitis B surface antigen, hepatitis C antibody screens;
  * Urinalysis: by dipstick; full microscopic examination if dipstick positive; and
  * Urine Drug Screen: ethyl alcohol, amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine metabolites, opiates, and phencyclidine.
  * Serum Pregnancy Screen (female subjects only)
  * FSH (to verify postmenopausal status; female subjects only)
* If female and:

  * is postmenopausal for at least 1 year and has a serum FSH level ≥ 20mIU/mL; or
  * is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).

Exclusion Criteria:

* Subjects with a recent history of dug or alcohol addiction or abuse.
* subjects with the presence of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease (as determined by the clinical investigators).
* Subjects whose clinical laboratory test values are outside the accepted reference range and when confirmed on re-examination are deemed to be clinically significant.
* Subjects demonstrating a reactive screen for hepatitis B surface antigen, hepatitis C antibody or HIV antibody.
* Subjects demonstrating positive drug abuse screen when screened for this study.
* Female subjects demonstrating a positive pregnancy screen.
* Female subjects who are currently breast-feeding.
* Subjects with a history of allergic response(s) to alprazolam or related drugs.
* Subjects with a history of clinically significant allergies including drug allergies.
* Subjects with a clinically significant illness during the 4 weeks prior to Period I dosing (as determined by the clinical investigators).
* Subjects who currently use or report using tobacco products within 90 days of Period I dose administration.
* Subjects who have taken any drug known to induce or inhibit hepatic drug metabolism in the 28 days prior to Period I dosing.
* Subjects who report donating greater than 150 mL of blood within 30 days prior to Period I dosing. All subjects will be advised not to donate plasma for four weeks after completing the study.
* Subjects who report receiving any investigational drug within 28 days prior to Period I dosing.
* Subjects who report taking any systemic prescription medication in the 14 days prior to Period I dosing.
* Subjects who report an intolerance of direct venipuncture.
* Subjects who report consuming an abnormal diet during the 28 days prior to Period I dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2005-06; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D. Carlson, Pharm. D., Principal Investigator — PRACS Institute, Ltd.
Locations (2):
- United States (2):
  - PRACS Institute, Ltd., East Grand Forks, Minnesota
  - PRACS Institute, Ltd., Fargo, North Dakota

RESULTS

PARTICIPANT FLOW:
Groups:
- Alprazolam (Test) First: Alprazolam 3 mg ER Tablet (test) dosed in first period followed by Xanax XR® 3 mg Tablet (reference) dosed in second period
- Xanax® (Reference) First: Xanax XR® 3 mg Tablet (reference) dosed in first period followed by Alprazolam 3 mg Tablet (test) dosed in second period
Period: First Intervention
Arm/Group | Alprazolam (Test) First | Xanax® (Reference) First
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0
Period: Washout: 7 Days
Arm/Group | Alprazolam (Test) First | Xanax® (Reference) First
Started | 16 | 16
Completed | 15 | 16
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Intervention
Arm/Group | Alprazolam (Test) First | Xanax® (Reference) First
Started | 15 | 16
Completed | 15 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alprazolam (Test) First | Xanax® (Reference) First | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 13 | 15 | 28
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 15 | 12 | 27
  Black | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native American or Alaskan Native | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Concentration
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 72 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Alprazolam: Alprazolam 3 mg ER Tablet (test) dosed in either period
- Xanax®: Xanax XR® 3 mg Tablet (reference) dosed in either period
Arm/Group | Alprazolam | Xanax®
Number analyzed (Participants) | 31 | 31
ng/mL | 24.33 (5.37) | 23.62 (4.29)
Statistical Analysis 1: Comparison: Alprazolam vs Xanax®; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% Confidence Interval falls withi 80-125; Geometric Test/Ref Ratio x 100 = 102.56, 90% CI 2-sided [98.74 to 106.52] — Bioequivalence is established when 90% Confidence Interval falls withi 80-125

2. Primary Outcome: AUC0-inf - Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated)
Description: Bioequivalence based on AUC0-inf
Time Frame: Blood samples collected over 72 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Alprazolam | Xanax®
Number analyzed (Participants) | 31 | 31
ng*h/mL | 668.79 (250.55) | 725.34 (291.34)
Statistical Analysis 1: Comparison: Alprazolam vs Xanax®; Test type: Non-Inferiority or Equivalence — An analysis of variance (ANOVA) was performed on each of the pharmacokinetic parameters using SAS® software; Geometric Test/Ref Ratio x 100 = 92.88, 90% CI [90.34 to 95.48] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

3. Primary Outcome: AUC0-t - Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant)
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 72 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Alprazolam | Xanax®
Number analyzed (Participants) | 31 | 31
ng*h/mL | 620.40 (213.87) | 663.08 (226.97)
Statistical Analysis 1: Comparison: Alprazolam vs Xanax®; Test type: Non-Inferiority or Equivalence — An analysis of variance (ANOVA) was performed on each of the pharmacokinetic parameters using SAS® software; Geometric Test/Ref Ratio x 100 = 93.92, 90% CI [91.47 to 96.44] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.